CLINICAL TRIAL: NCT01288079
Title: A Phase IIb, Randomized, Double-Blind, Placebo-Controlled, Active Controlled, Parallel Group, Multicenter Study to Assess the Safety and Efficacy of 2 Fixed Dose Groups of TC-5214 (S-mecamylamine) as Monotherapy Treatment in Patients With Major Depressive Disorder Who Exhibit an Inadequate Response to Antidepressant Therapy
Brief Title: A Study to Assess the Safety and Effect of TC-5214 in Patients With Major Depressive Disorder.
Status: Terminated | Phase: Phase 2 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: D4131C00001
Record Dates: First submitted 2011-01-26; First posted 2011-02-02 (Estimated); Results first posted 2012-10-29 (Estimated); Last update posted 2012-11-20 (Estimated); Status verified 2012-11

CONDITIONS: Major Depressive Disorder
Keywords: Major Depressive Disorder; MDD; Monotherapy; Inadequate Response to Antidepressant Therapy
MeSH Terms: conditions — Depressive Disorder, Major | interventions — Duloxetine Hydrochloride

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- 1 (Experimental): TC-5214, 1 mg BID
  Interventions: Drug: TC-5214
- 2 (Experimental): TC-5214, 4 mg BID
  Interventions: Drug: TC-5214
- 3 (Active Comparator): Duloxetine 60 mg Q Day
  Interventions: Drug: Duloxetine
- 4 (Placebo Comparator): Placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: TC-5214 — Tablet, oral, twice daily for 8 weeks
  Arms: 1; 2
Drug: Duloxetine — Capsule, oral, once daily
  Arms: 3
Drug: Placebo — Tablet, oral, twice daily for 8 weeks
  Arms: 4

SUMMARY:
The purpose of this study is to assess the safety and effect of TC-5214 as a single therapy in patients with major depressive disorder who exhibit inadequate response to antidepressants.

ELIGIBILITY:
Inclusion Criteria:

* Provision of signed and dated informed consent before initiation of any study-related procedures.
* The patient must have a clinical diagnosis of major depressive disorder (MDD) with inadequate response to no more than one antidepressant.
* Women of child-bearing potential must have a negative urine pregnancy test and confirmed use of a highly effective form of birth control before enrollment and until 3 months after their last dose of study drug.
* Outpatient status at enrollment and randomization.

Exclusion Criteria:

* Patients with a lifetime history of bipolar disorder; psychotic disorder or post-traumatic stress disorder.
* Patients with a history of suicide attempts in the past year and/or seen by the investigator as having a significant history of risk of suicide or homicide.
* Patients with any significant unstable hepatic, renal, pulmonary, cardiovascular, ophthalmologic, neurologic, or any other medical conditions that might confound the study or put the patient at greater risk during study participation.
* History of stroke or transient ischemic attack, seizures or seizure disorder, head trauma including closed head injury.
* Pregnancy or lactation.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 145 (Actual)
Dates: Start 2011-02; Primary Completion 2012-08 (Actual); Study Completion 2012-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Hans A Eriksson, MD, PhD, MBA, Study Director — AstraZeneca R&D Södertälje
Locations (63):
- United States (25):
  - Research Site, Beverly Hills, California
  - Research Site, Chino, California
  - Research Site, Garden Grove, California
  - Research Site, San Diego, California
  - Research Site, Torrance, California
  - Research Site, Bradenton, Florida
  - Research Site, Coral Springs, Florida
  - Research Site, Jacksonville, Florida
  - Research Site, North Miami, Florida
  - Research Site, St. Petersburg, Florida
  - Research Site, West Palm Beach, Florida
  - Research Site, Atlanta, Georgia
  - Research Site, Joliet, Illinois
  - Research Site, Prairie Village, Kansas
  - Research Site, Flowood, Mississippi
  - Research Site, New York, New York
  - Research Site, Rochester, New York
  - Research Site, Dayton, Ohio
  - Research Site, Mason, Ohio
  - Research Site, Portland, Oregon
  - Research Site, Allentown, Pennsylvania
  - Research Site, Dallas, Texas
  - Research Site, Houston, Texas
  - Research Site, Seattle, Washington
  - Research Site, Madison, Wisconsin
- Estonia (2):
  - Research Site, Tallinn
  - Research Site, Tartu
- Finland (4):
  - Research Site, Helsinki
  - Research Site, Jyväskylä
  - Research Site, Kuopio
  - Research Site, Tampere
- India (11):
  - Research Site, Visakhapatnam, Andh Prad
  - Research Site, Ahmedabad, Gujarat
  - Research Site, Bangalore, Kamataka
  - Research Site, Bangalore, Karnataka
  - Research Site, Mangalore, Karnataka
  - Research Site, Nashik, Mahara
  - Research Site, Jaipur, Rajasthan
  - Research Site, Chennai, Tamil Nadu
  - Research Site, Varanasi, Uttar Prad
  - Research Site, Kanpur
  - Research Site, Pune
- Japan (21):
  - Research Site, Nagoya, Aichi-ken
  - Research Site, Ichikawa, Chiba
  - Research Site, Noda, Chiba
  - Research Site, Fukuoka, Fukuoka
  - Research Site, Omuta, Fukuoka
  - Research Site, Sapporo, Hokkaido
  - Research Site, Sapproro, Hokkaido
  - Research Site, Akashi, Hyōgo
  - Research Site, Kobe, Hyōgo
  - Research Site, Kawasaki-shi, Kanagawa
  - Research Site, Sagamihara-shi, Kanagawa
  - Research Site, Yokohama, Kanagawa
  - Research Site, Kumamoto, Kumamoto
  - Research Site, Yatsushiro, Kumamoto
  - Research Site, Ukyo-ku ,Kyoto, Kyoto
  - Research Site, Kurashiki-shi, Okayama-ken
  - Research Site, Kodaira-shi, Tokyo
  - Research Site, Meguro-ku, Tokyo
  - Research Site, Minato-ku, Tokyo
  - Research Site, Setagaya-ku, Tokyo
  - Research Site, Shinagawa-ku, Tokyo

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This multicenter study was conducted in Europe, Asia, and North America between 4 February 2011 and 26 April 2012.
Pre-assignment Details: 21-day screening/washout and 8-week prospective open-label SSRI(selective serotonin reuptake inhibitors)/SNRI(selective serotonin and norepinephrine reuptake inhibitors) periods to identify population of inadequate responders(<50% reduction in Hamilton Rating Scale for Depression total score of ≥16 and a Clinical Global Impression-Severity ≥4).
Period: Overall Study
Arm/Group | 1 mg BID TC-5214 | 4 mg BID TC-5214 | 60 mg QD Duloxetine | Placebo
Started | 37 | 36 | 37 | 35
Completed | 17 | 9 | 18 | 18
Not Completed | 20 | 27 | 19 | 17
Not completed — Withdrawal by Subject | 2 | 4 | 1 | 0
Not completed — Adverse Event | 2 | 1 | 2 | 3
Not completed — Severe Non-Compliance to Protocol | 1 | 3 | 1 | 3
Not completed — Condition under Investigation Worsened | 0 | 0 | 0 | 1
Not completed — Lack of Efficacy | 2 | 2 | 0 | 2
Not completed — Study-Specific Withdrawal Criteria | 1 | 1 | 0 | 0
Not completed — Lost to Follow-up | 1 | 1 | 1 | 0
Not completed — Other or Study Termination | 11 | 15 | 14 | 8

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | 1 mg BID TC-5214 | 4 mg BID TC-5214 | 60 mg QD Duloxetine | Placebo | Total
Number analyzed (Participants) | 37 | 36 | 37 | 35 | 145
Age Continuous [Mean (Standard Deviation); unit: years] | 44.5 (13.03) | 40.3 (12.50) | 41.8 (12.70) | 40.1 (10.49) | 41.7 (12.24)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 24 | 26 | 22 | 19 | 91
  Male | 13 | 10 | 15 | 16 | 54
Race/Ethnicity, Customized [Number; unit: participants]
  White | 23 | 20 | 23 | 20 | 86
  Black or African American | 1 | 4 | 4 | 5 | 14
  Asian | 12 | 10 | 9 | 9 | 40
  Native Hawaiian or other Pacific Islander | 0 | 0 | 0 | 0 | 0
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Other | 1 | 2 | 1 | 1 | 5
Hamilton Rating Scale for Depression-17 items (HAMD-17) total score at randomization [Mean (Standard Deviation); unit: Scores on a scale] — A 17-item, clinician-rated scale that assesses depressive symptoms. The Hamilton Rating Scale for Depression-17 items (HAMD-17) consists of 17 symptoms, each of which is rated from 0 to 2 or 0 to 4, where 0 is none/absent. Higher HAMD-17 scores indicate more severe depression.
  Scores on a scale | 20.914 (3.425) | 21.371 (3.606) | 21.857 (3.499) | 21.344 (4.100) | 21.372 (3.632)
Montgomery-Asberg Depression Rating Scale (MADRS) total score at randomization [Mean (Standard Deviation); unit: Scores on a scale] — A 10-item scale for the evaluation of depressive symptoms. Each Montgomery-Asberg Depression Rating Scale (MADRS) item is rated on a 0 to 6 scale. The MADRS total score is calculated as the sum of the 10 individual item scores; the total score can range from 0 to 60. Higher MADRS scores indicate higher levels of depressive symptoms.
  Scores on a scale | 27.228 (5.202) | 26.857 (5.542) | 28.600 (6.796) | 27.625 (5.320) | 27.577 (5.734)

OUTCOME MEASURES:

1. Primary Outcome: Change in the Montgomery Asberg Depression Rating Scale (MADRS) Total Score From Randomization to End of Treatment
Description: A 10-item scale for the evaluation of depressive symptoms. Each Montgomery Asberg Depression Rating Scale (MADRS) item is rated on a 0 to 6 scale. The MADRS total score is calculated as the sum of the 10 individual item scores; the total score can range from 0 to 60. Higher MADRS scores indicate higher levels of depressive symptoms.
Time Frame: Randomization (Week 8) to end of treatment (Week 16)
Population: Modified intent-to-treat analysis set including all randomized patients who received at least 1 dose of investigational product (TC-5214, duloxetine or placebo) and who had a randomization and at least 1 post-randomization MADRS total score.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | 1 mg BID TC-5214 | 4 mg BID TC-5214 | 60 mg QD Duloxetine | Placebo
Number analyzed (Participants) | 35 | 35 | 35 | 32
units on a scale | -9.1 (2.15) | -11.2 (2.56) | -11.4 (2.14) | -7.6 (2.19)
Statistical Analysis 1: Comparison: 1 mg BID TC-5214 vs Placebo; Mixed model repeated measures (MMRM) includes treatment, pooled center, visit, treatment by visit interaction, region, responsiveness, and region by responsiveness as explanatory variables and the randomization MADRS total score as a covariate. Treatment, visit treatment by visit interaction, region, responsiveness, and region by responsiveness are fixed effects in the model; pooled center is a random effect; Test type: Superiority or Other; p = 0.617, MMRM; LS mean = -1.5, 95% CI 2-sided [-7.35 to 4.39], Standard Error of Mean 2.95
Statistical Analysis 2: Comparison: 4 mg BID TC-5214 vs Placebo; Mixed model repeated measures (MMRM) includes treatment, pooled center, visit, treatment by visit interaction, region, responsiveness, and region by responsiveness as explanatory variables and the randomization MADRS total score as a covariate. Treatment, visit, treatment by visit interaction, region, responsiveness, and region by responsiveness are fixed effects in the model; pooled center is a random effect; Test type: Superiority or Other; p = 0.277, MMRM; LS mean = -3.6, 95% CI 2-sided [-10.06 to 2.91], Standard Error of Mean 3.26
Statistical Analysis 3: Comparison: 60 mg QD Duloxetine vs Placebo; [analysis description as in outcome 1, analysis 2]; Test type: Superiority or Other; p = 0.194, MMRM; LS mean = -3.9, 95% CI 2-sided [-9.72 to 2.00], Standard Error of Mean 2.95

ADVERSE EVENTS:
Arm/Group | 1 mg BID TC-5214 | 4 mg BID TC-5214 | 60 mg QD Duloxetine | Placebo
Serious Adverse Events (participants affected / at risk) | 1/37 | 0/35 | 0/37 | 1/35
Other Adverse Events (participants affected / at risk) | 22/37 | 27/35 | 21/37 | 24/35
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 1 mg BID TC-5214 (N=37) | 4 mg BID TC-5214 (N=35) | 60 mg QD Duloxetine (N=37) | Placebo (N=35)
Abdominal Pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Subcutaneous Abscess (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 1 mg BID TC-5214 (N=37) | 4 mg BID TC-5214 (N=35) | 60 mg QD Duloxetine (N=37) | Placebo (N=35)
Anaemia Megaloblastic (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Eosinophilia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Leukopenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Neutropenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Tinnitus (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Vision Blurred (Eye disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Eye Pain (Eye disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Visual Impairment (Eye disorders) | 0 (0) | 0 (0) | 1 (2) | 1 (1)
Constipation (Gastrointestinal disorders) | 0 (0) | 9 (9) | 2 (2) | 2 (2)
Nausea (Gastrointestinal disorders) | 4 (4) | 3 (3) | 7 (9) | 2 (2)
Diarrhoea (Gastrointestinal disorders) | 1 (1) | 3 (3) | 1 (1) | 3 (3)
Abdominal Pain (Gastrointestinal disorders) | 2 (2) | 2 (2) | 0 (0) | 1 (1)
Dry Mouth (Gastrointestinal disorders) | 0 (0) | 2 (2) | 1 (1) | 0 (0)
Abdominal Pain Upper (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (2)
Dental Caries (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dyspepsia (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (4)
Flatulence (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Toothache (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Asthenia (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Drug Withdrawal Syndrome (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Fatigue (General disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Feeling Abnormal (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Feeling Cold (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pyrexia (General disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Thirst (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hepatic Function Abnormal (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Seasonal Allergy (Immune system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Influenza (Infections and infestations) | 1 (1) | 1 (1) | 2 (2) | 4 (4)
Nasopharyngitis (Infections and infestations) | 3 (3) | 2 (2) | 0 (0) | 3 (3)
Urinary Tract Infection (Infections and infestations) | 0 (0) | 2 (3) | 1 (1) | 1 (1)
Bronchitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Gastroenteritis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hordeolum (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Tooth Infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Upper Respiratory Tract Infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Urethritis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Procedural Dizziness (Injury, poisoning and procedural complications) | 1 (4) | 0 (0) | 2 (5) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Limb Injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Blood Pressure Increased (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 2 (2)
Heart Rate Increased (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Weight Decreased (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Weight Increased (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Increased Appetite (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 3 (3)
Decreased Appetite (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Dyslipidaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Folate Deficiency (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Back Pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 3 (3) | 0 (0)
Pain In Extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (2) | 0 (0) | 0 (0)
Joint Swelling (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Muscle Spasms (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Neck Pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pain In Jaw (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 6 (6) | 4 (4) | 5 (8) | 6 (8)
Headache (Nervous system disorders) | 4 (5) | 6 (6) | 3 (8) | 5 (8)
Somnolence (Nervous system disorders) | 2 (2) | 1 (1) | 4 (5) | 0 (0)
Dizziness Postural (Nervous system disorders) | 1 (1) | 0 (0) | 1 (1) | 3 (8)
Balance Disorder (Nervous system disorders) | 0 (0) | 0 (0) | 2 (2) | 1 (3)
Paraesthesia (Nervous system disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Disturbance In Attention (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dysgeusia (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Formication (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Head Discomfort (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Hypoaesthesia (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Memory Impairment (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Stupor (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Tremor (Nervous system disorders) | 1 (1) | 1 (1) | 1 (1) | 1 (1)
Insomnia (Psychiatric disorders) | 0 (0) | 3 (3) | 4 (4) | 2 (2)
Agitation (Psychiatric disorders) | 0 (0) | 1 (1) | 1 (1) | 2 (2)
Nightmare (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 2 (2)
Suicidal Ideation (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Abnormal Dreams (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Anxiety (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Bradyphrenia (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Confusional State (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dissociation (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hypervigilance (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Intentional Self-Injury (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Libido Decreased (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Mood Swings (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Sleep Disorder (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Tension (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Nocturia (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pollakiuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Urinary Retention (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Uterine Polyp (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 2 (2) | 1 (1) | 1 (1) | 0 (0)
Night Sweats (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Urticaria (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hypertension (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Orthostatic Hypotension (Vascular disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Varicose Vein (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)

LIMITATIONS AND CAVEATS:
The study was terminated early and thus only a fraction of the planned number of patients were randomized and many did not complete the study. As a consequence the possibility of interpreting efficacy over an 8 week period is considerably reduced.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days